CLINICAL TRIAL: NCT01573715
Title: Effects of NMBA on the Alteration of Transpulmonary Pressures at the Early Phase of ARDS
Brief Title: Effects of Neuromuscular Blocking Agents (NMBA) on the Alteration of Transpulmonary Pressures at the Early Phase of Acute Respiratory Distress Syndrome (ARDS)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-005720-18; 2011-39 (Other: AP HM)
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — cisatracurium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- severe ARDS patients (Active Comparator)
  Interventions: Drug: NIMBEX
- control group (Active Comparator)
  Interventions: Drug: NIMBEX; Other: WITHOUT NIMBEX
- moderate SDRA patients (Experimental)
  Interventions: Drug: NIMBEX; Other: WITHOUT NIMBEX

INTERVENTIONS:
Drug: NIMBEX
  Arms: severe ARDS patients
Drug: NIMBEX
  Arms: control group; moderate SDRA patients
Other: WITHOUT NIMBEX
  Arms: control group; moderate SDRA patients

SUMMARY:
Mortality in Acute Respiratory Distress Syndrome is high (40 to 60 %). Protective mechanical ventilation, until 2010, was the cornerstone of the ARDS therapeutic strategies. Recently, a prospective multicenter study demonstrates that a 48h continuous infusion of neuromuscular blocking agents (NMBA) have a positive impact on mortality of ARDS patients. (Papazian et al. ACURASYS Study. NEJM 2010; 363:1107-16). The mechanisms through which NMBAs could improve survival remain speculative. They are as follows:

* reduction of the consumption of oxygen linked to ventilatory workload;
* increase of chest wall compliance improving mechanical ventilation during ARDS and better adaptation to the protective ventilation strategy;
* anti-inﬂammatory effect contributing to a reduction in pulmonary inﬂammation and improvement in oxygenation,
* reduction of the variations of transpulmonary pressure (TPP) by the way of better synchronisation between patient and the ventilator.

The use of NMBA could also reduce the ventilator induced lung injury by a better control of TPP.

ELIGIBILITY:
Inclusion Criteria:

* Early (< 48H) Severe ARDS: PaO2 / FiO2 ratio < 150 with PEEP >= 5 cmH20

Exclusion Criteria:

Age < 18 ans Patient already under continuous infusion NMBA. Known NMBA Allergy or intolerance Contra-indication to introduction of nasogastric tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Delta TPP | 27 months
  Reduction of Delta TPP at 48 hr in the NMBA group by comparison with the control group in ARDS patients

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France